CLINICAL TRIAL: NCT03544983
Title: A Randomized Trial of Proactive Outreach and Streamlined Genetic Education in BRCA Families
Brief Title: Genetic Education in BRCA Families
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: George Washington University (Other)
Responsible Party: Principal Investigator, Marc D Schwartz, Professor of Oncology, Associate Director for Population Science, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2018-0439
Record Dates: First submitted 2018-05-22; First posted 2018-06-04 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: BRCA1 Mutation; BRCA2 Mutation
Keywords: Breast Cancer; Ovarian Cancer; Prostate Cancer; BRCA1; BRCA2
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Two group parallel design comparing Web-based education + streamlined telephone genetic information session to usual care.
Who Masked: Outcomes Assessor
Masking Description: Outcomes will be assessed via electronic survey and review of medical records. In cases where surveys need to be completed by telephone, the outcomes assessor will be blind to the participant's randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proactive Outreach + Web Counseling (Experimental): Web + Streamlined Telephone Genetic Information
  Interventions: Behavioral: Web + Streamlined Telephone Genetic Information
- Usual Care (No Intervention): Participants in the usual care arm will not be provided with access to the web-based intervention nor will they have access to streamlined genetic counseling. They can pursue clinical genetic counseling on their own.

INTERVENTIONS:
Behavioral: Web + Streamlined Telephone Genetic Information — Tailored and interactive web-based education designed to incorporate all aspects of standard genetic counseling followed by a streamlined genetic counseling session with a board-certified genetic counselor.
  Arms: Proactive Outreach + Web Counseling

SUMMARY:
The primary goal of this research is to test a web-based genetic education intervention that is designed to educate men and women from hereditary cancer families about the personal relevance of genetic testing in order to help them male decisions about whether to pursue genetic testing. We will test this intervention against standard care for men and women from hereditary cancer families. The web-based educational intervention includes all of the information typically covered during genetic counseling. As a result, after completing the education intervention, participants can proceed directly to a brief telephone call with a genetic counselor followed by testing if they choose. A baseline survey will be administered prior to randomization and then follow-up surveys will be administered at 1-month and 6-months post-randomization. Primary outcomes will be completion of genetic counseling, uptake of genetic testing, genetic test results and quality of life.

DETAILED DESCRIPTION:
Women who carry a pathogenic BRCA variant (PV) have a lifetime breast cancer risk of 55-70% and a lifetime ovarian cancer risk of 16-45%. Men with a PV are at increased risk for prostate, pancreatic and breast cancer. BRCA testing typically begins with a family member (proband) who is affected with cancer. If a PV is identified, probands are encouraged to communicate this test result with at risk relatives. Unaffected first- and second-degree relatives (FSDR), who are at 50% and 25% risk for carrying the PV, may then pursue genetic counseling and testing for the specific variant identified in the proband (targeted testing). Targeted testing is far less complex and expensive than testing probands and definitively distinguishes carriers from non-carriers. Such testing allows carriers to reduce their cancer incidence, morbidity and mortality through risk reduction and screening while non-carriers can avoid unnecessary medical intervention and their offspring can safely forgo testing. Despite these well-recognized significant benefits and clear guideline-based recommendations for genetic counseling and testing, only 28-57% of FSDRs undergo BRCA testing. This low rate of participation occurs despite high rates of result communication by probands, calling into question the quality of the information communicated and the accuracy of FSDRs understanding of the importance of the information. Additional barriers to counseling and testing include: limited access, lack of referral, time and travel commitment, and lack of proactive clinical approaches to facilitate uptake.

Remarkably, there have been no randomized trials focused on increasing use of guideline consistent genetic counseling and targeted testing. Guided by the Informed Choice (ICM) and Health Belief Models (HBM), the investigators will conduct a randomized controlled trial of proactive Web-based pre-test education plus a streamlined telephone genetic information session (W+T) vs usual care (UC) for unaffected FSDRs of PV carriers. Web-based pre-counseling education followed by a streamlined telephone genetic information session will be proactively delivered. Following counseling, participants will have the option to proceed directly to targeted testing. By proactively providing access to accurate genetic information and reducing barriers to genetic services, W+T is predicted to yield increased uptake of genetic counseling and testing.

Aim 1: Evaluate the impact of web-based intervention plus brief telephone information (W+T) vs. Usual Care (UC) on uptake of genetic counseling and targeted genetic testing.

Aim 2: Evaluate the impact of W+T vs UC on psychosocial outcomes.

Aim 3: Evaluate mechanisms and moderators of W+T.

Research Overview. The aim of this RCT is to evaluate the efficacy of proactively delivered Web Pre-Test Education plus Streamlined Telephone Counseling (W+T) for first- and second-degree relatives (FSDRs) of individuals who have recently received a positive BRCA test result (i.e., probands). The W+T intervention is designed to facilitate access to genetic education and counseling, foster informed decisions and reduce barriers to targeted genetic testing. The primary hypotheses are that W+T participants will have increased uptake of genetic counseling and targeted genetic testing relative to UC participants. Eligible FSDRs will be contacted for a baseline assessment. One-month following the baseline assessment, all participating FSDRs will be randomized (by family) to either W+T or UC. FSDRs will be reassessed at 1- and 6-months post-randomization and probands will be reassessed at 6-months post-randomization to enumerate additional testing in the family.

Identification and Enrollment. Probands will be recruited within the clinical genetics programs at LCCC, George Washington University (GWU), Geisinger Clinic, and Dana Farber Cancer Institute (DFCI); through direct referrals from local cancer genetics programs (MedStar Franklin Square Medical Center, Sibley Hospital, and Inova Schar Cancer Institute). We will enroll probands who have received a positive BRCA test result within the prior 12-months. At GLCCC and GWU we routinely obtain permission to recontact BRCA probands at the time of their test result disclosure. At Geisinger Clinic and DFCI, study staff will obtain and document participant permission to share contact information with the study team. For participants referred by outside clinical providers (Franklin Square, Sibley, and Inova), the provider will obtain patient permission to share contact information with the study team. We will also enroll self-referred probands who will be identified in two ways. First, we will advertise the study on social media (Facebook/Instagram/Google). Facebook/Instagram/Google users who click on the study advertisement will be taken to our study website where they can review basic study information or find contact information to reach the study team with any questions. Those who wish to proceed can then go directly to our secure REDCap page where they can complete a brief eligibility screener. Second, we will recruit self-referred probands who receive positive test results from the Ambry Genetics genetic testing laboratory. Patients who have received a positive BRCA1/BRCA2 test result within the past 12-months through Ambry will be identified by Ambry Genetics. Ambry Genetics will then provide study information to the ordering providers who will be asked to pass this information along wit a study invitation to their potentially eligible patients. Patients who respond to the study invitation will then be taken to the REDCap screening page described above. Eligible probands will be contacted for enrollment a minimum of one-month following disclosure and a maximum of 12-months. At that time they will be asked for consent to access their genetic counseling/testing records and provide the names, addresses, and telephone numbers of all potentially eligible FSDRs. Participating probands will be asked to inform all potentially eligible FSDRs about the planned study contact.

After obtaining contact information, potentially eligible FSDRs will be mailed a recruitment packet (introductory letter, study brochure, informed consent document, opt-out e-mail/address/telephone number). Two weeks later, a research assistant will call all FSDRs who have not opted out of the study. The RA will explain the study and answer any questions. At enrollment participants will be informed that written consent is required prior to randomization. They will also be informed of the randomization date and that they must complete their baseline survey before that date in order to participate in the study.

Baseline Assessment. Individuals who remain eligible and interested can complete the 20 minute baseline survey via telephone by a trained RA or electronically. For those who do not return the consent document prior to the baseline, an RA will use an IRB-approved verbal consent for telephone baselines or electronic consent for electronic baselines. Written consent will be required prior to randomization.

Randomization. Following the baseline, participants will be provided with a randomization date on which they will be contacted with their assignment. Participants will be randomized by family to avoid contamination. Randomization will take place 1 month after enrollment of the first FSDR in a family. At that point, FSDRs who have not completed a baseline will be ineligible for the study. Participants will be informed of the randomization deadline upon enrollment. On the randomization date, participants will be notified by email or phone, followed by a priority letter. For W+T participants, this letter will contain log-in information website instructions. For UC participants, this letter will include a list of informational resources (including a list of low-cost genetic counseling options).

Interventions.

Usual Care. As part of standard clinical genetic counseling, probands with a BRCA mutation are provided with an individualized summary letter that includes cancer risks, management recommendations and options, a family letter that identifies at-risk relatives and encourages them to share the test result with these relatives. All participants in both arms will receive these standard materials. As described above, following randomization, UC participants will be notified of their assignment and will receive a list of informational resources. Of course, they can pursue standard clinical genetic counseling on their own at any of our study sites or any other program.

The W+T Intervention. The W+T intervention includes: Interactive Pre-Test Web-Education plus a streamlined telephone information session (directly scheduled through the web site); and for those who opt for testing, a telephone genetic counseling disclosure session. The W+T pre-test Web component is designed to provide comparable information to a traditional genetic counseling session for an FSDR of a mutation carrier. A detailed description of the content of the W+T is described in the treatment plan below. Participants will receive an individualized link to the website that is connected to their email address. They will be able to create their own password the first time they access the website, and then log back into the website in the future using their email address and created password. The website has a "forgot password" option, where participants can create a new password at any time. The study will provide participants with a toll-free support number to call if they have any questions. After reviewing the website, participants will be provided with the option to schedule a brief telephone information session with a trained genetic research assistant. This session will take approximately 15 minutes and is designed to supplement and reinforce the web-based information. This session will be provided free of charge. Participants can decline

Genetic Testing. Genetic testing is not required as part of this study. Any participants who proceed with genetic testing will receive standard clinical testing for their familial mutation (or more extensive testing when clinically indicated). At the conclusion of the pre-test telephone counseling session, participants who wish to proceed directly to testing will have the process for testing explained by the genetic counselor and a test requisition form (TRF) including insurance information will be completed. Upon completion of the TRF, a DNA saliva collection kit will be sent via overnight mail to the participant. After participants collect their DNA, they mail the kit and all included paperwork to the lab in a pre-paid FedEx pack. Targeted testing will be for the specific PV identified in their family, and if Ashkenazi Jewish (AJ), also for the 3 BRCA founder mutations. In rare instances participants may have a particularly complex family history and will be appropriate for broader multiplex testing. This option will be explained by the genetic counselor during the telephone session.

Telephone Genetic Counseling Disclosure. Telephone disclosures will be delivered by the same board certified genetic counselors who provided pretest counseling. Telephone disclosures will utilize our existing clinical disclosure protocol that includes: result disclosure with comprehensive interpretation; discussion of cancer risks and management options; implications for family members; referral to specialists as needed/indicated. Within a week of the disclosure session, participants will be provided with a copy of their results, pedigree and an individualized summary letter.

Follow-Up Survey. Participants will be contacted for follow-up surveys at 1-month and 6-months post-randomization. These surveys will be similar to (but shorter than) the baseline survey.

ELIGIBILITY:
Inclusion Criteria:

* A first- (sibling, adult offspring) or second-degree (aunt/uncle, niece/nephew if at-risk parent is deceased) biological relative of an individual with a recently identified BRCA1 or BRCA2 mutation

Exclusion Criteria:

* Personal diagnosis of metastatic cancer
* Prior genetic testing for hereditary breast/ovarian cancer
* Have one or more children who have tested positive for a BRCA1 or BRCA2 mutation
* Cannot participate in or understand English
* Cannot provide meaningful informed consent

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Uptake of genetic counseling and testing | 6-months post randomization
  The proportion of participants who complete genetic counseling and testing

SECONDARY OUTCOMES:
Patient Reported Outcomes Measurement Information System -- Anxiety | 1- and 6-months post-randomization
  Measures anxiety symptoms. Scores are calculated as T-Scores with a mean of 50 and a standard deviation of 10. Higher scores indicate more anxiety.
Patient Reported Outcomes Measurement Information System -- Depression | 1- and 6-months post-randomization
  Measures depression symptoms. Scores are calculated as T-Scores with a mean of 50 and a standard deviation of 10. Higher scores indicate more depression.
Decisional Conflict Scale | 1- and 6-months post-randomization
  The decisional conflict scale (DCS) measures personal perceptions of: a) uncertainty in choosing between medical options; b) modifiable factors contributing to uncertainty such as feeling uninformed, unclear about personal values and unsupported in decision making; and c) effective decision making such as feeling the choice is informed, values-based, likely to be implemented and expressing satisfaction with the choice.
  The scale consists of 16-items each with 5 response categories. Subscales are: 1) informed subscale; 2) values clarity subscale; 3) support subscale; 4) uncertainty subscale; 5) effective decision subscale. The total score is calculated by taking the average item score across all 16 items and multiplying by 25 to yield a range of 0 - 100 in which higher scores indicate greater decisional conflict.
Multidimensional Impact of Cancer Risk Scale - Uncertainty Scale | 6-months post-randomization
  The uncertainty subscale of the Multidimensional Impact of Cancer Risk scale consists of 9-items that are summed to create a final uncertainty score. Higher scores indicate greater concerns regarding the uncertainty of genetic test results.

CONTACTS AND LOCATIONS:
Overall Officials: Marc D Schwartz, PhD, Principal Investigator — Georgetown University
Locations (4):
- United States (4):
  - Georgetown University Medical Center/Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - George Washington University, Washington D.C., District of Columbia
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Geisinger Medical Center, Danville, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
We do not plan to share IPD with other researchers.